CLINICAL TRIAL: NCT03715231
Title: NIDEK Gonioscope GS-1 for Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-00429
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glaucoma & Glaucoma Suspect Patients (Experimental): Patients with Glaucomatous optic neuropathy
  Interventions: Other: NIDEK Gonioscope GS-1; Other: Standard Digital Gonioscopic Images

INTERVENTIONS:
Other: NIDEK Gonioscope GS-1 — To determine inter-observer repeatability when using this device, two observers will examine each image obtained from NIDEK Gonioscope GS-1 and separately determine the iridocorneal angle. Inter-observer repeatability will be tested using Pearson correlation.
Other: Standard Digital Gonioscopic Images — To determine inter-observer repeatability when using this device, two observers will examine each image obtained from NIDEK Gonioscope GS-1 and separately determine the iridocorneal angle. Inter-observer repeatability will be tested using Pearson correlation.

SUMMARY:
The Gonioscope GS-1 is an ophthalmic camera with gonioscopic prism that is intended to capture, display and store images of the anterior chamber angle and its peripheral part. This study evaluates the efficiency of Gonioscope GS-1 in glaucoma patients.With the captured images, the glaucoma diagnosis and post-operative observation are enabled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with glaucoma or glaucoma suspect

Glaucoma Suspect

* Glaucomatous optic neuropathy as described in the glaucoma patients below
* AND/OR ocular hypertension (IOP > 21 mm Hg)
* Normal visual field

Glaucoma Patients

* Clinical characteristics of glaucoma: ONH abnormalities: global rim thinning, rim notch, or disc hemorrhage; RNFL defect
* Typical glaucomatous field loss in reliable VF, reproducible glaucoma hemifield tests labeled outside normal limits on at least two consecutive tests.
* Both eyes will be included, except in cases where only one eye meets study criteria

Exclusion Criteria:

* Corneal opacities (scars, edema, etc.)
* Pregnant or planning to become pregnant
* Inability to fixate gaze

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Inter-Observer Repeatability for NIDEK Gonioscope GS-1 | 1 Day
  To determine reliability, two observers will examine images from NIDEK Gonioscopes GS-1. Repeatability will mean observations of both observers will coincide.
Inter-Observer Repeatability for Standard Digital Gonioscopic images | 1 Day
  To determine reliability, two observers will examine images from NIDEK Gonioscopes GS-1. Repeatability will mean observations of both observers will coincide.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Schuman, Principal Investigator — NYUMC Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). To achieve aims in the approved proposal.Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Requests should be directed to Zena.Moore@nyulangone.org to gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Madu CT, Phelps T, Schuman JS, Zambrano R, Lee TF, Panarelli J, Al-Aswad L, Wollstein G. Automated 360-degree goniophotography with the NIDEK Gonioscope GS-1 for glaucoma. PLoS One. 2023 Mar 7;18(3):e0270941. doi: 10.1371/journal.pone.0270941. eCollection 2023. PMID 36881575